CLINICAL TRIAL: NCT05693610
Title: Comparing Outcomes With the Cloud-based and Portable Versions of an Open-source Hearing Aid.
Brief Title: Open-source Hearing Aid Platform Comparisons
Acronym: COSP-1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was paused after April 2023 as the decision was made to continue the study with an updated version of test devices. However, the devices are still in production and the site is being closed for the study due to relocation of the PI.
Sponsor: Northwestern University (Other)
Collaborators: Nadi LLC (Industry)
Responsible Party: Principal Investigator, Varsha Rallapalli, Research Assistant Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Pro00062688
Record Dates: First submitted 2022-06-08; First posted 2023-01-23 (Actual); Results first posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: Hearing Loss; Hearing Loss, Sensorineural
Keywords: Hearing aid; Hearing loss
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: Within-subjects design; Different levels of intervention outcomes are compared
Masking Description: Since the portable and cloud-based versions of the device are visibly different, it is not possible to mask the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Portable OSP (Experimental): Outcomes will be assessed with the portable version of the OSP.
  Interventions: Device: Portable OSP
- Cloud-based OSP (Experimental): Outcomes will be assessed with the cloud-based version of the OSP.
  Interventions: Device: Cloud-based OSP

INTERVENTIONS:
Device: Portable OSP — The portable open-source speech processing platform (OSP) is accessed on a browser via a wireless fidelity (WiFi)-enabled portable communication device that carries out all the signal processing. The processed sounds are transmitted to the ears via earpieces known as behind-the-ear receivers in the canal (same as those available with commercial hearing aids). The amount of amplification with the portable OSP will be customized for each listener based on a validated prescription.
  Arms: Portable OSP
Device: Cloud-based OSP — The cloud-based open-source speech processing platform (OSP) is hosted on a web-server which includes the software for all the signal processing. The processed sounds are transmitted to the ears via calibrated headphones. The amount of amplification with the cloud-based OSP will be customized for each listener based on a validated prescription.
  Arms: Cloud-based OSP

SUMMARY:
New discoveries for hearing loss intervention are often impeded by the proprietary nature of commercial hearing aids and their use in scientific research as "black boxes". An open-source speech platform (OSP) was developed to bridge the gap between audiology research and commercial hearing aid features, to promote innovative solutions to meet the needs of the hearing loss community. The OSP can replicate functions found in commercial hearing aids, and provides tools to researchers to access those functions. The purpose of this study is to evaluate portable and cloud-based platforms of the OSP that will enable a wide range of lab and field applications. All human subjects-related activities will be conducted at Northwestern University (single-site study).

DETAILED DESCRIPTION:
New discoveries for hearing loss intervention are often impeded by the proprietary nature of commercial hearing aids and their use in scientific research as "black boxes". An open-source hearing aid (open-source speech platform or OSP) was developed to bridge the gap between audiology research and the commercialization of hearing aid technologies and to promote innovative solutions to meet the needs of the hearing loss community. The OSP can replicate functions found in commercial hearing aids, and provides tools to researchers and listeners to access those functions. The purpose of this study is to evaluate portable and cloud-based platforms of the OSP that will enable a wide range of lab and field applications by measuring speech perception abilities with the open-source hearing aid in quiet and in noise for adults with and without hearing loss.

The study is a within-subjects design that allows for the comparison of outcomes within the same participant. The study will compare performance with two platforms of the open-source hearing aid (portable and cloud-based) for adults with hearing loss and normal hearing. The study will measure performance using tests of word identification. We will test aided performance with clinically validated hearing aid settings in quiet and in noise. Each participant will be presented with all the test conditions, and the order of presentation of the test conditions will be randomized across participants. Statistical analyses will use a repeated measures model to control for correlation between outcomes for the same participant.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age; any sex
* Sensorineural hearing loss with pure-tone thresholds between 25-85 decibel hearing level (dB HL) at octave frequencies between 250 and 3000 Hz
* Speak English as their primary language
* Normal or corrected-to-normal vision
* Participants will be in good health (self-report)

Exclusion Criteria:

* Clinically significant unstable or progressive medical conditions
* Participants who score < 23 on the cognitive screening test (Montreal Cognitive Assessment)
* Evidence of conductive hearing loss or middle ear issues
* Significant history of otologic or neurologic disorders
* Non English-speaking or non-native English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Varsha H Rallapalli, AuD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a single arm, within-subjects study design and each participant completed both study interventions. First the portable OSP was tested followed by the cloud-based OSP for all participants.
Groups:
- Portable OSP, Then Cloud-based OSP: Outcomes will be assessed with the portable and cloud-based versions of the OSP.
  Portable OSP: The portable open-source speech processing platform (OSP) is accessed on a browser via a wireless fidelity (WiFi)-enabled portable communication device that carries out all the signal processing. The processed sounds are transmitted to the ears via earpieces known as behind-the-ear receivers in the canal (same as those available with commercial hearing aids). The amount of amplification with the portable OSP will be customized for each listener based on a validated prescription.
  Cloud-based OSP: The cloud-based open-source speech processing platform (OSP) is hosted on a web-server which includes the software for all the signal processing. The processed sounds are transmitted to the ears via calibrated headphones. The amount of amplification with the cloud-based OSP will be customized for each listener based on a validated prescription.
Period: Overall Study
Arm/Group | Portable OSP, Then Cloud-based OSP
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Portable OSP, Then Cloud-based OSP
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (23.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Word-identification Ability
Description: Word identification ability will be assessed using the Modified Rhyme Test. Participants will select a word out of a choice of six rhyming words. The words may be in quiet or mixed with background noise and will be presented through headphones (for the intervention type: cloud-based OSP) or via loudspeakers (for the intervention type: portable OSP). Participants may be asked to record their responses on paper or via a button/mouse click on a computer or tablet screen. Scores will be based on the percentage of words identified correctly (range: 0-100%). A higher score indicates better word identification ability. The task is expected to take 30 minutes for each test condition.
Time Frame: Post-intervention (1 day)
Population: Includes individuals with normal hearing and hearing loss
Measure: Mean (95% Confidence Interval); unit: percentage of words correct
Arm/Group | Portable OSP | Cloud-based OSP
Number analyzed (Participants) | 11 | 11
percentage of words correct | 78.12 [71.54 to 84.71] | 85.07 [80.77 to 89.36]

2. Secondary Outcome: Phoneme Confusions
Description: Phoneme confusions will be obtained from the Modified Rhyme Test conducted in outcome measure 1. The phoneme confusions will be derived by comparing the selected words to the target word in the task and will be presented in terms of number or percentage of substitution, insertion, deletion errors. No addition task is required for this outcome measure.
Time Frame: Post-intervention (1 day)
Population: Due to errors in the software, this outcome measure was not collected for any of the participants.
Arm/Group | Portable OSP, Then Cloud-based OSP
Number analyzed (Participants) | 0

3. Secondary Outcome: Response Time
Description: Response time will be obtained from the Modified Rhyme Test conducted in outcome measure 1. Response time is a measure of time taken (in seconds) to identify a word correctly or incorrectly.
Time Frame: Post-intervention (1 day)
Population: Includes individuals with normal hearing and hearing loss.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Portable OSP | Cloud-based OSP
Number analyzed (Participants) | 11 | 10
seconds | 3.91 [3.51 to 4.30] | 3.60 [3.27 to 3.94]

ADVERSE EVENTS:
Time Frame: No adverse events to report because all-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Portable OSP | Cloud-based OSP
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2024-03-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT05693610/Prot_SAP_000.pdf
  • Informed Consent Form: Main Consent Form (2024-03-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT05693610/ICF_001.pdf
  • Informed Consent Form: Screener Consent Form (2024-03-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT05693610/ICF_002.pdf